CLINICAL TRIAL: NCT04284579
Title: Determination Effective Dose 95 (ED95) of Intravenous Cannulation With the Induction of Sevoflurane 8 Vol% in Patients Aged 1-3 Years Using Dixon up and Down Method
Brief Title: Optimum Time for Intravenous Cannulation After Induction With Sevoflurane in Pediatric Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Jefferson K Hidayat, MD, Indonesia University
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IndonesiaUAnes50
Record Dates: First submitted 2020-02-23; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Movement After Intravenous Cannulation
Keywords: child, general anesthesia, induction of anesthesia, sevoflurane, venous cannulation
MeSH Terms: interventions — Cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- time for cannulation (Experimental): intravenous cannulation after sevoflurane induction
  Interventions: Device: IV cannula

INTERVENTIONS:
Device: IV cannula — We measure the time duration needed for IV cannulation

SUMMARY:
This study aimed to determinate effective dose 95 (ED95) intravenous cannulation in pediatric patient after induction of sevoflurane 8 vol%

DETAILED DESCRIPTION:
Twenty-two subjects were given informed consent before study enrolled. Anesthesia was induced by 8% sevoflurane with 6 L flow of 100% oxygen. IV cannulation was attempted at 2 min in the first child in each group. The time for cannulation in the next child was stepped up or down by 15 s depending on positive or negative response, respectively, in the previous child. Children were recruited till a minimum of six pairs of failure-success sequence which was obtained in the group. The mean of midpoints of the failure-success sequence was calculated to obtain the time for cannulation in 50% of the group.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-3 year
* Physical state ASA I dan II
* Parents of patients who agreed to participate and sign informed consent.

Exclusion criteria:

* Patients with difficult airway
* There's allergic reaction or drug's side effect after induction
* There's cardiorespiratory problem such as anaphylactic shock, aritmia, severe hypotension, desaturation before-on-or after induction

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
ED50 in intravenous cannulation after sevoflurane induction | 2 minutes
  using Dixon Up and Down Method

CONTACTS AND LOCATIONS:
Overall Officials: Jefferson K Hidayat, Principal Investigator — Indonesia University
Locations (1):
- Indonesia University, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schwartz D, Connelly NR, Gutta S, Freeman K, Gibson C. Early intravenous cannulation in children during sevoflurane induction. Paediatr Anaesth. 2004 Oct;14(10):820-4. doi: 10.1111/j.1460-9592.2004.01315.x. PMID 15385009
- [Result] Kumar KR, Sinha R, Chandiran R, Pandey RK, Darlong V, Chandralekha. Evaluation of optimum time for intravenous cannulation after sevoflurane induction of anesthesia in different pediatric age groups. J Anaesthesiol Clin Pharmacol. 2017 Jul-Sep;33(3):371-374. doi: 10.4103/joacp.JOACP_58_16. PMID 29109638
- [Result] Kilicaslan A, Gok F, Erol A, Okesli S, Sarkilar G, Otelcioglu S. Response to Makkar and Singh's comment on our article 'Determination of optimum time for intravenous cannulation after induction with sevoflurane and nitrous oxide in children premedicated with midazolam'. Paediatr Anaesth. 2015 Mar;25(3):328-9. doi: 10.1111/pan.12611. No abstract available. PMID 25623378
- [Result] Whalen FX, Bacon DR, Smith HM. Inhaled anesthetics: an historical overview. Best Pract Res Clin Anaesthesiol. 2005 Sep;19(3):323-30. doi: 10.1016/j.bpa.2005.02.001. PMID 16013684
- [Result] Behne M, Wilke HJ, Harder S. Clinical pharmacokinetics of sevoflurane. Clin Pharmacokinet. 1999 Jan;36(1):13-26. doi: 10.2165/00003088-199936010-00002. PMID 9989340